CLINICAL TRIAL: NCT04955847
Title: Efficacy and Safety of Oral Misoprostol 25 μg vs. Vaginal Dinoprostone in Induction of Labor at Term
Acronym: MISODINO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0070
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Induction of Labor; Vaginal Delivery; Cesarean Section
Keywords: Induction of Labor; PGE1; PGE2; vaginal delivery; cesarean section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PGE2: In period 1, the service protocol for induction at term on an unfavorable cervix indicated the use of a PGE2. In nulliparous women, Propess® was introduced intra-vaginally for 24 hours or until regular painful uterine contractions occurred. In the case of a multiparous woman, Prostine® gel, one or two mg depending on the cervical conditions at the time of induction, was introduced intravaginally and the cervix was reassessed after six hours. If the cervix remained unfavorable and the kinetics of the contractions were not optimal, a new dose of Prostine® one or two mg was administered to the patient.
- misoprostol: In period 2, patients who were induced with an unfavorable cervix at term were induced with misoprostol. Regardless of parity, the patient received oral misoprostol 25 μg, one tablet orally every two hours until a maximum of eight tablets per day, or 200 µg, was reached, with cessation of the tablets when painful, regular contractions were obtained.

SUMMARY:
Labor induction is a common medical technique. There is no consensus on which technique is better than the others. Misoprostol is an analogue of Prostaglandin E1 previously used off-label in labor induction. Its low cost, room-temperature storage, and diverse route options have made it an alternative to PGE2 in labor induction. As of 2018, oral misoprostol 25 μg tablet was licensed for labor induction.

Very few studies have been performed on oral misoprostol 25 μg and none compared it with the PGE2s mostly used in induction on unfavorable cervix at term.

The investigators compared the safety and the efficacy between the oral misoprostol 25 μg Angusta® used since 20/02/2020 and the vaginal dinoprostone previously used in gel or diffuser over two consecutive periods from 01/01/2019 to 19/02/2020 for the dinoprostone and from 20/02/2020 to 07/04/2021 for the misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* age of patient> 18 years
* patients requiring induction of labor with a singleton pregnancy at term, a gestational age greater than 37 weeks of amenorrhea, with a fetus in cephalic presentation and an unfavorable cervix (Bishop score less than six).

Exclusion Criteria:

* intrauterine fetal death,
* preterm pregnancy,
* scarred uterus
* contraindications to vaginal delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: all patients requiring induction of labor with a singleton pregnancy at term, a gestational age greater than 37 weeks of amenorrhea, with a fetus in cephalic presentation and an unfavorable cervix (Bishop score less than six)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Variation of vaginal deliveries within 24hours patient number in both groups | 24 hours

SECONDARY OUTCOMES:
Variation of Cesarean section patient number in both groups | 24 hours
Variation of indications for cesarean section in both groups | 24 hours
Variation of uterine contractility abnormalities in both groups | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No